CLINICAL TRIAL: NCT06258031
Title: PsilOCD: Evaluating the Effects of the 5-HT2A Agonist Psilocybin on the Neurocognitive and Clinical Correlates of Compulsivity (A Pharmacological-Challenge Feasibility Study)
Brief Title: PsilOCD: A Pharmacological-Challenge Feasibility Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 298206
Record Dates: First submitted 2024-01-08; First posted 2024-02-14 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Two different, fixed doses of psilocybin (Dose A = 10mg - x, Dose B = 10mg - y) are given on two separate dosing days to all patients.
Masking Description: Study is single group, but participants are blinded to the fixed doses received on both dosing days (Dose A and Dose B), and the outcomes assessor responsible for evaluating OCD and depression symptoms using the Y-BOCS and MADRS is also blinded. Assessors evaluating all other outcomes are unblinded.
  Note to editor: I ticked 'None (Open Label)' as advised, to avoid this being flagged and to be able to release this protocol; it is impossible to accurately describe our study's design with these options available. Please may this 'None (Open Label)' description be removed once it is published?
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All participants (Experimental): Up to 10mg of psilocybin on two separate dosing days (separated by 4 weeks)
  Interventions: Drug: Psilocybin (COMP360)

INTERVENTIONS:
Drug: Psilocybin (COMP360) — Up to 10mg on two occasions
  Other Names: O-phosphoryl-4-hydroxy-N,N-dimethyltryptamine

SUMMARY:
The purpose of this study is to assess the impact of psilocybin on cognitive inflexibility and neural plasticity in a cohort of people with obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
This mechanistic study will utilise a within-subjects design, administering up to 10mg of psilocybin to participants with OCD (DSM-5 criteria) on two separate instances spaced four weeks apart. To ensure consistency and participant safety, dosing will occur under medical supervision with psychological support from two experienced therapists. Before and after each session, participants will engage in virtual preparation and integration sessions led by their therapists. Cognitive tasks will be administered in the days following each dosing session. Additionally, acute post-dosing EEG recordings will be conducted, and blood samples will be taken after each dosing session. OCD symptoms will also be assessed seven times throughout the trial by an external blinded psychiatrist, serving as a secondary outcome. Collectively, these measures aim to evaluate changes in cognitive inflexibility, decision-making abilities, neuroplasticity (peripheral blood markers and EEG measures), inflammation (peripheral blood markers), and symptomatology following each dosing session.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 20 to 65 years;
* Any gender;
* A primary diagnosis of OCD (based on the Mini-International Neuropsychiatric Interview (M.I.N.I.));
* Has met diagnostic criteria for OCD for at least 12 months;
* Willing to comply with protocol and associated lifestyle restrictions;
* Adequate understanding of the English language to give informed consent and participate in the study;
* Participant can attend visits as an outpatient;
* Comfortable using a computer, access to internet from home, and willing to participate in some of the study visits via video-link.

Key Exclusion Criteria:

* Current or past history of dependent (according to ICD10 criteria) substance use (not including nicotine and/or caffeine), Tourette's syndrome, autism spectrum disorder, epilepsy, organic mental disorder, or a personality disorder apart from obsessive-compulsive personality disorder;
* Current or past history of psychosis or mania in themselves or a first-degree relative;
* Unstable physical health;
* Significantly abnormal clinical test result;
* Heavy smoker, or unable to attend the dosing days (including the subsequent recovery part) without a smoking break;
* Unwillingness to allow their GP or mental health practitioners to be informed of their participation (or, to allow study team access to Summary Care Record).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Intradimensional-extradimensional (ID-ED) set shift | 4 weeks
  Scores on this neurocognitive task administered as part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). ID-ED performance is an established measure of cognitive inflexibility in OCD (Chamberlain et al., Am J Psychiatry, 2007), with worse scores corresponding to decreased flexibility.
The visual long-term potentiation (vLTP) electroencephalogram (EEG) paradigm (acute quantified changes in neuroplasticity in the visual system). | 8 weeks
  We will assess acute changes in homosynaptic neuroplasticity using the visual long-term potentiation (vLYTP) EEG paradigm. In this paradigm, we induce neural plasticity in the occipital cortex by exposing participants to visual stimuli of varying frequencies. This task specifically quantifies homosynaptic plasticity because it triggers changes in neighbouring neurons within the occipital cortex.

SECONDARY OUTCOMES:
Clinical measures of compulsivity of relevance to OCD including Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 8 weeks
  Assess OCD symptoms over the study's duration (with higher scores corresponding to worse symptoms in all scales mentioned)
Cognitive measure: Reversal learning task (administered as part of the Cambridge Neuropsychological Test Automated Battery (CANTAB)) | 4 weeks
  Assesses ability to adapt to changing contingencies; higher scores indicate better cognitive flexibility
Cognitive measure: Information-seeking task | 4 weeks
  It tests participants' confidence and ability to make decisions involving uncertainty by monitoring their tendency to seek extra information (recently developed by Lion Schulz and colleagues, 2020)
Cognitive measure: Visuospatial memory paired-associates learning task (administered as part of the Cambridge Neuropsychological Test Automated Battery (CANTAB)) | 4 weeks
  Serves as a control task; higher scores indicate better visuospatial memory faculties
Measures of the acute psychological effects of psilocybin including the Emotional Breakthrough Inventory | 4 weeks
  Higher scores correspond to greater subjective emotional changes elicited by the acute psilocybin experience
Measures of depression symptoms including the Montgomery-Åsberg Depression Rating Scale (MADRS) | 8 weeks
  Higher scores correspond to worse depressive symptoms
Measures of anxiety symptoms including the State-Trait Anxiety Inventory (STAI) | 8 weeks
  Higher scores correspond to worse anxiety-related symptoms
Acute plasma serum concentration of Brain-Derived Neurotrophic Factor (BDNF) | 4 weeks
  BDNF concentration (pg/mL) serves as a biomarker with significant functions in brain health, neuroplasticity, and the regulation of inflammation.
Oura: heart-rate variability | 8 weeks
  Participants will be given an Oura ring to keep track of heart-rate variability (HRV) throughout the duration of the study (participants will not be able to see their own data).
Oura: sleep stages | 8 weeks
  Oura rings will also measure the number of minutes/hours spent in each sleep stage (awake, light, deep, and rapid eye movement (REM))
Oura: REM sleep | 4 weeks
  Examines acute changes in neuroplasticity. Participants detect subtle colour changes while listening to sound sequences, triggering an EEG signal increase in the auditory cortex. This measures the brain's ability to induce repetition suppression across consecutive trials, reflecting its capacity to adapt to expected sound sequences over time.

CONTACTS AND LOCATIONS:
Overall Officials: Professor David Nutt, Principal Investigator — Imperial College London; Dr David Erritzoe, Principal Investigator — Imperial College London; Dr Luca Pellegrini, Principal Investigator — University of Hertfordshire/Imperial College London; Professor Naomi Fineberg, Principal Investigator — University of Hertfordshire
Locations (1):
- CIPPRes Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No